CLINICAL TRIAL: NCT02706028
Title: Effects of Underwater Ultrasound Therapy on Hand Function and Quality of Life in Patients With Rheumatoid Arthritis - a Randomized Controlled Study
Brief Title: Effects of Underwater Ultrasound Therapy on Hand Function and Quality of Life in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petz Aladar County Teaching Hospital (Other)
Responsible Party: Principal Investigator, Márta Király, chief physician, Petz Aladar County Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PetzACTH
Record Dates: First submitted 2016-02-29; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
Keywords: underwater ultrasound; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound group (Active Comparator): Patients in the ultrasound group received underwater US therapy to both hands and wrists for 7 minutes with an intensity of 0.7 W/cm2 in a total of 10 sessions (10 working days) using a 830 kHz ULTRON home OE-302® device with treatment head size of 4.2 cm2.
  Interventions: Device: underwater ultrasound
- control group (Sham Comparator): The control group received sham treatment (the ULTRON home OE-302® device was not turned on) during 10 sessions for 7 minutes per session.
  Interventions: Device: sham underwater ultrasound

INTERVENTIONS:
Device: underwater ultrasound — underwater US therapy with an intensity of 0.7 W/cm2 in a total of 10 sessions (10 working days) using a 830 kHz ULTRON home OE-302® device with treatment head size of 4.2 cm2.
  Arms: ultrasound group
Device: sham underwater ultrasound — ULTRON home OE-302® device is not turned on
  Arms: control group

SUMMARY:
In this randomized, double-blind, placebo-controlled study the effects of underwater ultrasound (US) therapy were investigated in 48 patients with moderately active rheumatoid arthritis (disease activity score in 28 joints (DAS28) ≥3.2 and ≤5.1).

Patients randomly assigned to the ultrasound group (N=25) received underwater ultrasound therapy to both wrists and hands for 7 minutes per session with an intensity of 0.7 W/cm2 during 10 sessions. The control group (N=23) received sham treatment under the same conditions. At baseline, at the end of treatment (Week 2) and at the follow-up visit (Week 14), the following parameters were evaluated: disease activity - erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), tender and swollen joint counts, pain on a visual analogue scale, and DAS28, hand function (fist making, wrist extension and flexion, hand grip strength), quality of life - Health Assessment Questionnaire (HAQ), and the patients rated their own condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with mild-to-moderate (DAS28 > 3.2 and < 5.1) rheumatoid arthritis meeting the American College of Rheumatology (ACR) diagnostic criteria
* No distinction was made between seropositive and seronegative patients (regarding rheumatoid factor and anti-citrullinated peptide antibody)
* a stable-dose pharmacotherapy (DMARDs therapy), NSAIDs, steroid) given for at least 2 months
* no physiotherapy within 1 month before starting the study

Exclusion Criteria:

* included high disease activity (DAS28 > 5.1) and remission (DAS28 < 2.6)
* other concomitant autoimmune diseases
* stable-dose pharmacotherapy for less than 2 months
* conditions contraindicating US therapy (severe osteoporosis when T-score < -3.5; infection; fever; osteomyelitis; pregnancy; untreated high blood pressure)
* physiotherapy within 1 month before starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
change in erythrocyte sedimentation rate | week 0 and week 2
  change from baseline erythrocyte sedimentation rate (ESR) at Week 2
change in erythrocyte sedimentation rate | week 0 and week 14
  change from baseline erythrocyte sedimentation rate (ESR) at Week 14
change in C-reactive protein | week 0 and week 2
  change from baseline C-reactive protein (CRP) at Week 2
change in C-reactive protein | week 0 and week 14
  change from baseline C-reactive protein (CRP) at Week 14
change in disease activity | week 0 and week 2
  change from baseline disease activity score (DAS28) at week 2
change in disease activity | week 0 and week 14
  change from baseline disease activity score (DAS28) at week 14
change in number of painful and swollen joints | week 0 and week 2
  change from baseline number of painful and swollen joints at week 2
change in number of painful and swollen joints | week 0 and week 14
  change from baseline number of painful and swollen joints at week 14
change in severity of pain at rest | week 0 and week 2
  change from baseline severity of pain at rest recorded on a 10 cm visual analogue scale (VAS) at week2
change in severity of pain at rest | week 0 and week 14
  change from baseline severity of pain at rest recorded on a 10 cm visual analogue scale (VAS) at week 14
change in duration of morning stiffness | week 0 and week2
  change from baseline duration of morning joint stiffness (minutes) at Week 2
change in duration of morning stiffness | week 0 nd week 14
  change from baseline duration of morning joint stiffness (minutes) at Week 14

SECONDARY OUTCOMES:
change in joint function (range of motion of the wrist) | week 0 and week 2
  change from baseline range of motion in the wrists (degrees) at week 2
change in joint function (range of motion of the wrist) | week 0 and week 14
  change from baseline range of motion in the wrists (degrees) at week 14
change in degree of fist making | week 0 and week 2
  change from baseline degree of fist making (based on nail tilting, 3 grades were used: 0: insufficient, 1: incomplete, 2: complete) at week 2
change in degree of fist making | week 0 and week14
  change from baseline degree of fist making (based on nail tilting, 3 grades were used: 0: insufficient, 1: incomplete, 2: complete) at week 2
change in hand grip strength | week 0 and week 2
  change from baseline hand grip strength (kg) at week 2
change in hand grip strength | week 0 and week 14
  change from baseline hand grip strength (kg) at week 14
change in quality of life | week 0 and week 2
  change from baseline quality of life (Health Assessment Questionnaire (HAQ) at week 2
change from baseline quality of life | week 0 and week 14
  change from baseline quality of life (Health Assessment Questionnaire (HAQ) at week 14

CONTACTS AND LOCATIONS:
Locations (1):
- Petz Aladár County Teaching Hospital, Győr, Válassza Ki A Megyét, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiraly M, Varga Z, Szanyo F, Kiss R, Hodosi K, Bender T. Effects of underwater ultrasound therapy on pain, inflammation, hand function and quality of life in patients with rheumatoid arthritis - a randomized controlled trial. Braz J Phys Ther. 2017 May-Jun;21(3):199-205. doi: 10.1016/j.bjpt.2017.04.002. Epub 2017 Apr 13. PMID 28442212